CLINICAL TRIAL: NCT00538954
Title: A Randomised Controlled Trial of Optimised Surgical Recovery: the Potential Synergy Between Enhanced Gastrointestinal Motility and Oral Nutritional/ Metabolic Support
Brief Title: Optimised Recovery With Accelerated Nutrition and GI Enhancement
Acronym: ORANGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: UEdinburgh
Record Dates: First submitted 2007-10-02; First posted 2007-10-03 (Estimated); Last update posted 2010-11-05 (Estimated); Status verified 2007-10

CONDITIONS: Colorectal Liver Metastases
Keywords: Perioperative; recovery; nutrition; enhanced; laxative
MeSH Terms: interventions — Magnesium Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): Follow a standard Enhanced Recovery After Surgery protocol
  Interventions: Other: Standard ERAS group
- 2 (Experimental): Follow a standard Enhanced Recovery After Surgery protocol and will receive 1 g of Magnesium Oxide laxative twice daily from the day after surgery until discharge
  Interventions: Drug: Post operative laxation (Magnesium Oxide)
- 3 (Experimental): Follow a standard Enhanced Recovery After Surgery protocol and will receive preconditioning with carbohydrate and fluid loading prior to surgery (800ml of Nutricia Preop the evening before surgery and 400 the morning of surgery 2 hours prior to anaesthesia) and postoperative nutritional supplements (200 ml Nutricia Fortisip twice daily) after surgery for 30 days
  Interventions: Dietary Supplement: Preoperative metabolic conditioning postoperative nutritional supplementation
- 4 (Experimental): Follow a standard Enhanced Recovery After Surgery protocol and will receive preconditioning with carbohydrate and fluid loading prior to surgery (800ml of Nutricia Preop the evening before surgery and 400 the morning of surgery 2 hours prior to anaesthesia) and postoperative nutritional supplements (200 ml Nutricia Fortisip twice daily) after surgery for 30 days and will receive postoperative laxative in the form of 20 ml of Magnesium Oxide twice daily form the day after surgery until discharge
  Interventions: Drug: Post operative laxation (Magnesium Oxide); Dietary Supplement: Preoperative metabolic conditioning postoperative nutritional supplementation

INTERVENTIONS:
Drug: Post operative laxation (Magnesium Oxide) — 20 ml of Magnesium Oxide twice daily from the day after surgery until discharge
  Arms: 2; 4
Dietary Supplement: Preoperative metabolic conditioning postoperative nutritional supplementation — Nutricia PreOP drinks 800 ml between 8-10 pm the evening before surgery Nutricia PreOP drinks 400 ml completed 2 hours before anaesthesia on the morning of surgery Nutricia Fortisip drinks 2 x 200 ml drinks from the day after surgery until day 30
  Arms: 3; 4
Other: Standard ERAS group
  Arms: 1

SUMMARY:
Factors which delay recovery following uncomplicated abdominal surgery include uncontrolled pain, intolerance of diet and poor mobility. Enhanced recovery after Surgery (ERAS) programmes are perioperative care pathways that address systematically these issues (i.e. improved dynamic pain relief, optimised nutritional care and enforced mobilisation) to promote a faster recovery and a shorter stay. The key treatments that improve outcome within an ERAS programme are not known. Moreover there are few acceptable, objective endpoints to assess key outcome variables such as return of GI function. This randomised trial will assess the potential synergy between early recovery of GI function (laxation) and early postoperative oral nutritional support(with associated preoperative preconditioning using carbohydrate/fluid loading). The main overall outcome targets being improved recovery of gastrointestinal function, postoperative nutritional status and physical function. It will validate the use of a novel, objective technique to measure gastric motility (surrogate for GI function). Such refinement of ERAS should result in shorter hospital stay and better use of limited health care resource.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing hepatic resection for benign or malignant conditions
* Able to understand the nature of the study and what will be required of them.
* Men and non-pregnant, non-lactating women
* BMI 18 - 30

Exclusion Criteria:

* Inability to give written, informed consent
* Patients with dementia or neurological impairment
* Patients with pre-existing condition limiting mobility
* Planned bile duct excision
* Repeat or staged procedures
* Central extended resections
* Underlying cirrhotic liver disease
* Jaundice (Bilirubin > 50 μmol/L)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2006-08; Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Recovery of gastrointestinal function: Time to pass flatus/stool (hours following the end of surgery) | Number of hours post surgery

SECONDARY OUTCOMES:
t ½ Gastric emptying time on the morning of post-operative day 3 | Postoperative day 3
Length of hospital stay: nights spent in hospital post-op | Until discharge
Patient activity level: measured by activPAL® activity meter | postoperative day 2 - 7 and day 30 - 37

CONTACTS AND LOCATIONS:
Overall Officials: Paul Hendry, MBChB, Principal Investigator — University of Edinburgh
Locations (2):
- University Hospital Maastricht, Maastricht, Netherlands
- Edinburgh Royal Infirmary, Edinburgh, United Kingdom

REFERENCES:
- [Derived] Hendry PO, van Dam RM, Bukkems SF, McKeown DW, Parks RW, Preston T, Dejong CH, Garden OJ, Fearon KC; Enhanced Recovery After Surgery (ERAS) Group. Randomized clinical trial of laxatives and oral nutritional supplements within an enhanced recovery after surgery protocol following liver resection. Br J Surg. 2010 Aug;97(8):1198-206. doi: 10.1002/bjs.7120. PMID 20602497